CLINICAL TRIAL: NCT02184273
Title: Randomized, Double Blind, Comparative Trial of the Efficacy and Tolerability of Nolotil i.v. vs. Placebo i.v. in the Prevention of Postoperative Pain in Children of 6 and 11 Years Old Undergoing Minor Surgery
Brief Title: Efficacy and Tolerability of Nolotil i.v. vs. Placebo i.v. in the Prevention of Postoperative Pain in Children Undergoing Minor Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1093.18
Record Dates: First submitted 2014-07-08; First posted 2014-07-09 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — metamizole magnesium

ARMS (2):
- Magnesium metamizol (Experimental)
  Interventions: Drug: Magnesium metamizol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium metamizol
  Other Names: Nolotil
  Arms: Magnesium metamizol
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to assess the analgesic efficacy in the prevention of postoperative pain in children undergoing minor surgery (herniorraphy, tonsillectomy) and to assess the tolerability of Metamizol in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Children of either sex between 6 and 11 years of age
* Patients undergoing routine inguinal hernia repair or tonsillectomy
* Written informed consents by the guardian, according to the guidelines of Good Clinical Practice and current legislation
* The ability of the patient to understand and carry out the visual analogue scale assessments
* Patients with a physical status American Society of Anesthesiologist I or II class

Exclusion Criteria:

* The use of any drug with analgesic properties in the 24 hours prior to the administration of the study drug
* Surgery with a foreseen duration over 60 minutes
* Patients with a nutritional index of less than 90 or greater than 120
* Patients with a body mass index which was not between the 3rd centile and the 97th centile for age
* Patients with any illness or malformation (except hernia) which, in the doctor's opinion, contraindicated the use of metamizol (aplastic anemia, agranulocytosis of a toxicological etiology, severe renal disease, etc.)
* Patients who have received in the previous 7 days or need currently anticoagulant treatment
* Significant allergy or known hypersensitivity to metamizol, its excipients and/or to other nonsteroidal antiinflammatory drugs
* Patients in whom the anesthetic regimen required by the protocol cannot be used
* Patients who have participated in another clinical trial in the past four weeks or are currently participating in another clinical trial
* Patients with any psychological disturbance which, in the investigator's opinion makes the patient unsuitable for inclusion in the trial

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2002-03; Primary Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Percentage of children requiring rescue medication | up to 4 hours after drug administration

SECONDARY OUTCOMES:
Time from drug administration, end of surgery and first patient's awake to the administration of rescue medication | up to 4 hours
Percentage of children who require rescue medication | up to 2 hours after drug administration
Evaluation of the pain intensity by the patient by means of a Visual Analogue Scale (VAS) | up to 4 hours
Evaluation of the pain intensity by the patient by means of a four points Verbal Rating Scale (VRS) | up to 4 hours
Assessment of the state of the patient by the guardian by means of the Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) test | up to 4 hours
Assessment of the partial efficacy by the investigator by means of a four points VRS | up to 4 hours
Assessment of the total efficacy by the investigator by means of a four points VRS | after 4 hours
Number of patients with adverse events (AE) | up to 4 hours
Number of withdrawals due to AEs | up to 4 hours
Assessment of the total tolerability of the assigned treatment by the investigator by means of a four points VRS | after 4 hours